CLINICAL TRIAL: NCT02503293
Title: A Randomised, Cross-over Study to Compare Quality of Life and Satisfaction in Primary Immunodeficient Patients Treated With Subcutaneous Injections of Gammanorm® 165 mg/mL Administered With Two Different Delivery Devices: Injections Using Pump or Rapid Push
Brief Title: A Study to Compare Quality of Life and Satisfaction in Primary Immunodeficient Patients Treated With Subcutaneous Injections of Gammanorm® 165 mg/mL Administered With Two Different Delivery Devices: Injections Using Pump or Rapid Push
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GAN-06
Record Dates: First submitted 2015-07-01; First posted 2015-07-20 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Primary Immunodeficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chrono Super PID then Generic Syringe - Gammanorm (Other): Each patient will receive the study treatment using each of the two studied delivery devices according to the sequence randomly assigned based on a cross-over design:
  • Chrono Super PID then Generic Syringe-Gammanorm
  Interventions: Device: Chrono Super PID then Generic Syringe-Gammanorm
- Generic Syringe then Chrono Super PID - Gammanorm (Other): Each patient will receive the study treatment using each of the two studied delivery devices according to the sequence randomly assigned based on a cross-over design:
  • Generic Syringe then Chrono Super PID-Gammanorm
  Interventions: Device: Generic Syringe then Chrono Super PID-Gammanorm

INTERVENTIONS:
Device: Chrono Super PID then Generic Syringe-Gammanorm — Each patient will receive the study treatment of Gammanorm using each of the two studied delivery devices according to the sequence randomly assigned based on a cross-over design:
  • pump and then syringe
  The use of automatic, programmable, compact pumps (such as CRONO SUPER PID) allows patients to remain mobile without interrupting their activities. Patients can infuse several sites simultaneously with infusion rates of up to 40 mL/h at 2 to 4 sites (abdomen, thighs, upper arms, lower back).
  Rapid and manual administration of SCIg using a syringe could therefore represent an alternative method by decreasing the duration of administration (around 10 minutes per injection at 1 or 2 sites simultaneously). The injection is self-administered by the patient. The infusion rate usually is 1 to 2 mL/min. The use of low viscosity products could facilitate injection
  Other Names: Automatic Programable compact pump - Chrono Super PID Pump
  Arms: Chrono Super PID then Generic Syringe - Gammanorm
Device: Generic Syringe then Chrono Super PID-Gammanorm — Each patient will receive the study treatment using each of the two studied delivery devices according to the sequence randomly assigned based on a cross-over design:
  • syringe and then pump.
  The use of automatic, programmable, compact pumps (such as CRONO SUPER PID) allows patients to remain mobile without interrupting their activities. Patients can infuse several sites simultaneously with infusion rates of up to 40 mL/h at 2 to 4 sites (abdomen, thighs, upper arms, lower back).
  Rapid and manual administration of SCIg using a syringe could therefore represent an alternative method by decreasing the duration of administration (around 10 minutes per injection at 1 or 2 sites simultaneously). The injection is self-administered by the patient. The infusion rate usually is 1 to 2 mL/min. The use of low viscosity products could facilitate injection
  Other Names: Automatic Programable compact pump - Chrono Super PID Pump
  Arms: Generic Syringe then Chrono Super PID - Gammanorm

SUMMARY:
A randomised, cross-over study to compare quality of life and satisfaction in primary immunodeficient patients treated with subcutaneous injections of Gammanorm® 165 mg/mL administered with two different delivery devices: injections using pump or rapid push.

ELIGIBILITY:
Inclusion criteria:

* Adult patients (≥ 18 years).
* Presenting with primary immunodeficiency.
* Having received subcutaneous injections of immunoglobulin at home using an automatic pump or syringe for at least 1 month at the time of inclusion.
* For whom the investigator decides to maintain immunoglobulin replacement therapy with subcutaneous injections of Gammanorm® 165 mg/mL at home.
* Freely given written informed consent from patient.
* Women of childbearing potential must have a negative result on a pregnancy test (human chorionic gonadotropine [HCG]-based assay) and need to practice contraception using a method of proven reliability for the duration of the study.

Exclusion Criteria:

• Participating in another interventional clinical study and receiving investigational medicinal product within three months before study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-07-29 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
To compare satisfaction (LQI questionnaire, factor I: treatment interference) in PID patients receiving subcutaneous injections of Gammanorm® 165 mg/mL by delivery device used. | Participants will be followed for a total of 6 months
  Each patient will be treated for two consecutive periods of three months each according to the sequence assigned based on the cross-over design (syringe and then pump, or pump and then syringe) without any intermediate washout period. The total duration of study treatment will therefore be 6 months for each patient. Assessment will be conducted via the LQI scale.

SECONDARY OUTCOMES:
To compare the other quality of life scores | Participants will be followed for a total of 6 months
  Each patient will be treated for two consecutive periods of three months each according to the sequence assigned based on the cross-over design (syringe and then pump, or pump and then syringe) without any intermediate washout period. The total duration of study treatment will therefore be 6 months for each patient.
  Assessment will be conducted via the LQI scale factors II and III Patient quality of life will be assessed via SF-36 scale. Patient satisfaction will be assessed via TSQM-11 scale

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Warnatz, MD, Principal Investigator — Centre of Chronic Immunodeficiency, University Medical Centre Freiburg, Breisacher
Locations (12):
- Australia (2):
  - CampbelltownHospital, Campbelltown
  - Canberra Hospital, Canberra
- Germany (2):
  - University Medical Centre Freiburg, Freiburg im Breisgau
  - Municipal Hospital "St. Georg", Leipzig
- Italy (2):
  - Azienda Ospedaliera di Padova, Allergologia ed Immunologia Clinica, Padua
  - Policlinic Umberto I - Universita di Roma "Sapienza", Clinical Immunology, Rome
- United Kingdom (6):
  - University Hospitals Birmingham, Birmingham
  - University Hospital of Wales, Cardiff
  - - The Royal London Hospital, London
  - The Royal Free, London
  - John Radcliff Hospital, Oxford
  - Derriford Hospital, Plymouth

REFERENCES:
- [Background] Kobrynski L. Subcutaneous immunoglobulin therapy: a new option for patients with primary immunodeficiency diseases. Biologics. 2012;6:277-87. doi: 10.2147/BTT.S25188. Epub 2012 Aug 24. PMID 22956859
- [Background] Gardulf A. Immunoglobulin treatment for primary antibody deficiencies: advantages of the subcutaneous route. BioDrugs. 2007;21(2):105-16. doi: 10.2165/00063030-200721020-00005. PMID 17402794
- [Background] Al-Herz W, Bousfiha A, Casanova JL, Chapel H, Conley ME, Cunningham-Rundles C, Etzioni A, Fischer A, Franco JL, Geha RS, Hammarstrom L, Nonoyama S, Notarangelo LD, Ochs HD, Puck JM, Roifman CM, Seger R, Tang ML. Primary immunodeficiency diseases: an update on the classification from the international union of immunological societies expert committee for primary immunodeficiency. Front Immunol. 2011 Nov 8;2:54. doi: 10.3389/fimmu.2011.00054. eCollection 2011. PMID 22566844
- [Background] Al-Herz W, Bousfiha A, Casanova JL, Chatila T, Conley ME, Cunningham-Rundles C, Etzioni A, Franco JL, Gaspar HB, Holland SM, Klein C, Nonoyama S, Ochs HD, Oksenhendler E, Picard C, Puck JM, Sullivan K, Tang ML. Primary immunodeficiency diseases: an update on the classification from the international union of immunological societies expert committee for primary immunodeficiency. Front Immunol. 2014 Apr 22;5:162. doi: 10.3389/fimmu.2014.00162. eCollection 2014. PMID 24795713
- [Background] Gardulf A, Bjorvell H, Gustafson R, Hammarstrom L, Smith CI. The life situations of patients with primary antibody deficiency untreated or treated with subcutaneous gammaglobulin infusions. Clin Exp Immunol. 1993 May;92(2):200-4. doi: 10.1111/j.1365-2249.1993.tb03380.x. PMID 7683584
- [Background] Tcheurekdjian H, Palermo T, Hostoffer R. Quality of life in common variable immunodeficiency requiring intravenous immunoglobulin therapy. Ann Allergy Asthma Immunol. 2004 Aug;93(2):160-5. doi: 10.1016/S1081-1206(10)61469-X. PMID 15328676
- [Background] Gardulf A, Nicolay U, Asensio O, Bernatowska E, Bock A, Carvalho BC, Granert C, Haag S, Hernandez D, Kiessling P, Kus J, Pons J, Niehues T, Schmidt S, Schulze I, Borte M. Rapid subcutaneous IgG replacement therapy is effective and safe in children and adults with primary immunodeficiencies--a prospective, multi-national study. J Clin Immunol. 2006 Mar;26(2):177-85. doi: 10.1007/s10875-006-9002-x. Epub 2006 Apr 26. PMID 16758340
- [Background] Busse PJ, Razvi S, Cunningham-Rundles C. Efficacy of intravenous immunoglobulin in the prevention of pneumonia in patients with common variable immunodeficiency. J Allergy Clin Immunol. 2002 Jun;109(6):1001-4. doi: 10.1067/mai.2002.124999. PMID 12063531
- [Background] Liese JG, Wintergerst U, Tympner KD, Belohradsky BH. High- vs low-dose immunoglobulin therapy in the long-term treatment of X-linked agammaglobulinemia. Am J Dis Child. 1992 Mar;146(3):335-9. doi: 10.1001/archpedi.1992.02160150075025. PMID 1543181
- [Background] Nolte MT, Pirofsky B, Gerritz GA, Golding B. Intravenous immunoglobulin therapy for antibody deficiency. Clin Exp Immunol. 1979 May;36(2):237-43. PMID 477026
- [Background] Pourpak Z, Aghamohammadi A, Sedighipour L, Farhoudi A, Movahedi M, Gharagozlou M, Chavoshzadeh Z, Jadid L, Rezaei N, Moin M. Effect of regular intravenous immunoglobulin therapy on prevention of pneumonia in patients with common variable immunodeficiency. J Microbiol Immunol Infect. 2006 Apr;39(2):114-20. PMID 16604243
- [Background] Roifman CM, Lederman HM, Lavi S, Stein LD, Levison H, Gelfand EW. Benefit of intravenous IgG replacement in hypogammaglobulinemic patients with chronic sinopulmonary disease. Am J Med. 1985 Aug;79(2):171-4. doi: 10.1016/0002-9343(85)90006-3. PMID 4025374
- [Background] Winkelstein JA, Conley ME, James C, Howard V, Boyle J. Adults with X-linked agammaglobulinemia: impact of disease on daily lives, quality of life, educational and socioeconomic status, knowledge of inheritance, and reproductive attitudes. Medicine (Baltimore). 2008 Sep;87(5):253-258. doi: 10.1097/MD.0b013e318187ed81. PMID 18794707
- [Background] Gardulf A, Nicolay U. Replacement IgG therapy and self-therapy at home improve the health-related quality of life in patients with primary antibody deficiencies. Curr Opin Allergy Clin Immunol. 2006 Dec;6(6):434-42. doi: 10.1097/01.all.0000246619.49494.41. PMID 17088648
- [Background] Buckley RH, Schiff RI. The use of intravenous immune globulin in immunodeficiency diseases. N Engl J Med. 1991 Jul 11;325(2):110-7. doi: 10.1056/NEJM199107113250207. No abstract available. PMID 2052044
- [Background] Cherin P, Cabane J. Relevant criteria for selecting an intravenous immunoglobulin preparation for clinical use. BioDrugs. 2010 Aug 1;24(4):211-23. doi: 10.2165/11537660-000000000-00000. PMID 20623988
- [Background] Berger M. Subcutaneous immunoglobulin replacement in primary immunodeficiencies. Clin Immunol. 2004 Jul;112(1):1-7. doi: 10.1016/j.clim.2004.02.002. PMID 15207776
- [Background] Church JA, Leibl H, Stein MR, Melamed IR, Rubinstein A, Schneider LC, Wasserman RL, Pavlova BG, Birthistle K, Mancini M, Fritsch S, Patrone L, Moore-Perry K, Ehrlich HJ; US-PID-IGIV 10% -Study Group10. Efficacy, safety and tolerability of a new 10% liquid intravenous immune globulin [IGIV 10%] in patients with primary immunodeficiency. J Clin Immunol. 2006 Jul;26(4):388-95. doi: 10.1007/s10875-006-9025-3. Epub 2006 May 17. PMID 16705486
- [Background] Stein MR, Nelson RP, Church JA, Wasserman RL, Borte M, Vermylen C, Bichler J; IgPro10 in PID study group. Safety and efficacy of Privigen, a novel 10% liquid immunoglobulin preparation for intravenous use, in patients with primary immunodeficiencies. J Clin Immunol. 2009 Jan;29(1):137-44. doi: 10.1007/s10875-008-9231-2. Epub 2008 Sep 24. PMID 18814020
- [Background] Wasserman RL, Church JA, Stein M, Moy J, White M, Strausbaugh S, Schroeder H, Ballow M, Harris J, Melamed I, Elkayam D, Lumry W, Suez D, Rehman SM. Safety, efficacy and pharmacokinetics of a new 10% liquid intravenous immunoglobulin (IVIG) in patients with primary immunodeficiency. J Clin Immunol. 2012 Aug;32(4):663-9. doi: 10.1007/s10875-012-9656-5. Epub 2012 Mar 6. PMID 22392046
- [Background] Brennan VM, Salome-Bentley NJ, Chapel HM; Immunology Nurses Study. Prospective audit of adverse reactions occurring in 459 primary antibody-deficient patients receiving intravenous immunoglobulin. Clin Exp Immunol. 2003 Aug;133(2):247-51. doi: 10.1046/j.1365-2249.2003.02199.x. PMID 12869031
- [Background] Gardulf A, Moller G, Jonsson E. A comparison of the patient-borne costs of therapy with gamma globulin given at the hospital or at home. Int J Technol Assess Health Care. 1995 Spring;11(2):345-53. doi: 10.1017/s0266462300006942. PMID 7540602
- [Background] Waniewski J, Gardulf A, Hammarstrom L. Bioavailability of gamma-globulin after subcutaneous infusions in patients with common variable immunodeficiency. J Clin Immunol. 1994 Mar;14(2):90-7. doi: 10.1007/BF01541341. PMID 7515071
- [Background] Chapel HM, Spickett GP, Ericson D, Engl W, Eibl MM, Bjorkander J. The comparison of the efficacy and safety of intravenous versus subcutaneous immunoglobulin replacement therapy. J Clin Immunol. 2000 Mar;20(2):94-100. doi: 10.1023/a:1006678312925. PMID 10821460
- [Background] Fasth A, Nystrom J. Safety and efficacy of subcutaneous human immunoglobulin in children with primary immunodeficiency. Acta Paediatr. 2007 Oct;96(10):1474-8. doi: 10.1111/j.1651-2227.2007.00485.x. Epub 2007 Sep 10. PMID 17850391
- [Background] Berger M, Murphy E, Riley P, Bergman GE; VIRTUE Trial Investigators. Improved quality of life, immunoglobulin G levels, and infection rates in patients with primary immunodeficiency diseases during self-treatment with subcutaneous immunoglobulin G. South Med J. 2010 Sep;103(9):856-63. doi: 10.1097/SMJ.0b013e3181eba6ea. PMID 20689467
- [Background] Misbah S, Sturzenegger MH, Borte M, Shapiro RS, Wasserman RL, Berger M, Ochs HD. Subcutaneous immunoglobulin: opportunities and outlook. Clin Exp Immunol. 2009 Dec;158 Suppl 1(Suppl 1):51-9. doi: 10.1111/j.1365-2249.2009.04027.x. PMID 19883424
- [Background] Gardulf A, Hammarstrom L, Smith CI. Home treatment of hypogammaglobulinaemia with subcutaneous gammaglobulin by rapid infusion. Lancet. 1991 Jul 20;338(8760):162-6. doi: 10.1016/0140-6736(91)90147-h. PMID 1712881
- [Background] Gardulf A, Bjorvell H, Andersen V, Bjorkander J, Ericson D, Froland SS, Gustafson R, Hammarstrom L, Nystrom T, Soeberg B, et al. Lifelong treatment with gammaglobulin for primary antibody deficiencies: the patients' experiences of subcutaneous self-infusions and home therapy. J Adv Nurs. 1995 May;21(5):917-27. doi: 10.1046/j.1365-2648.1995.21050917.x. PMID 7541407
- [Background] Hagan JB, Fasano MB, Spector S, Wasserman RL, Melamed I, Rojavin MA, Zenker O, Orange JS. Efficacy and safety of a new 20% immunoglobulin preparation for subcutaneous administration, IgPro20, in patients with primary immunodeficiency. J Clin Immunol. 2010 Sep;30(5):734-45. doi: 10.1007/s10875-010-9423-4. Epub 2010 May 8. PMID 20454851
- [Background] Hansen S, Gustafson R, Smith CI, Gardulf A. Express subcutaneous IgG infusions: decreased time of delivery with maintained safety. Clin Immunol. 2002 Sep;104(3):237-41. doi: 10.1006/clim.2002.5215. PMID 12217333
- [Background] Gardulf A, Andersen V, Bjorkander J, Ericson D, Froland SS, Gustafson R, Hammarstrom L, Jacobsen MB, Jonsson E, Moller G, et al. Subcutaneous immunoglobulin replacement in patients with primary antibody deficiencies: safety and costs. Lancet. 1995 Feb 11;345(8946):365-9. doi: 10.1016/s0140-6736(95)90346-1. PMID 7845120
- [Background] Radinsky S, Bonagura VR. Subcutaneous immunoglobulin infusion as an alternative to intravenous immunoglobulin. J Allergy Clin Immunol. 2003 Sep;112(3):630-3. doi: 10.1016/s0091-6749(03)01781-0. No abstract available. PMID 13679829
- [Background] Gardulf A, Bjorvell H, Gustafson R, Hammarstrom L, Smith CI. Safety of rapid subcutaneous gammaglobulin infusions in patients with primary antibody deficiency. Immunodeficiency. 1993;4(1-4):81-4. No abstract available. PMID 7513227
- [Background] Nicolay U, Kiessling P, Berger M, Gupta S, Yel L, Roifman CM, Gardulf A, Eichmann F, Haag S, Massion C, Ochs HD. Health-related quality of life and treatment satisfaction in North American patients with primary immunedeficiency diseases receiving subcutaneous IgG self-infusions at home. J Clin Immunol. 2006 Jan;26(1):65-72. doi: 10.1007/s10875-006-8905-x. PMID 16418804
- [Background] Gardulf A, Nicolay U, Math D, Asensio O, Bernatowska E, Bock A, Costa-Carvalho BT, Granert C, Haag S, Hernandez D, Kiessling P, Kus J, Matamoros N, Niehues T, Schmidt S, Schulze I, Borte M. Children and adults with primary antibody deficiencies gain quality of life by subcutaneous IgG self-infusions at home. J Allergy Clin Immunol. 2004 Oct;114(4):936-42. doi: 10.1016/j.jaci.2004.06.053. PMID 15480339
- [Background] Kittner JM, Grimbacher B, Wulff W, Jager B, Schmidt RE. Patients' attitude to subcutaneous immunoglobulin substitution as home therapy. J Clin Immunol. 2006 Jul;26(4):400-5. doi: 10.1007/s10875-006-9031-5. Epub 2006 Jun 17. PMID 16783533
- [Background] Remvig L, Andersen V, Hansen NE, Karle H. Prophylactic effect of self-administered pump-driven subcutaneous IgG infusion in patients with antibody deficiency: a triple-blind cross-over study comparing P-IgG levels of 3 g l-1 versus 6 g l-1. J Intern Med. 1991 Jan;229(1):73-7. doi: 10.1111/j.1365-2796.1991.tb00309.x. PMID 1995766
- [Background] Long AA, Denburg JA, Dent PB. Hypogammaglobulinemia: therapeutic rationale. CMAJ. 1987 Nov 1;137(9):793-7. PMID 3327579
- [Background] Beaute J, Levy P, Millet V, Debre M, Dudoit Y, Le Mignot L, Tajahmady A, Thomas C, Suarez F, Pellier I, Hermine O, Aladjidi N, Mahlaoui N, Fischer A; French PID study group CEREDIH. Economic evaluation of immunoglobulin replacement in patients with primary antibody deficiencies. Clin Exp Immunol. 2010 May;160(2):240-5. doi: 10.1111/j.1365-2249.2009.04079.x. Epub 2009 Dec 16. PMID 20041884
- [Background] Shapiro R. Subcutaneous immunoglobulin therapy by rapid push is preferred to infusion by pump: a retrospective analysis. J Clin Immunol. 2010 Mar;30(2):301-7. doi: 10.1007/s10875-009-9352-2. Epub 2010 Jan 15. PMID 20082124
- [Background] Hogy B, Keinecke HO, Borte M. Pharmacoeconomic evaluation of immunoglobulin treatment in patients with antibody deficiencies from the perspective of the German statutory health insurance. Eur J Health Econ. 2005 Mar;6(1):24-9. doi: 10.1007/s10198-004-0250-5. PMID 15480920
- [Background] Haddad L, Perrinet M, Parent D, Leroy-Cotteau A, Toguyeni E, Condette-Wojtasik G, Hachulla E. [Economic evaluation of at home subcutaneous and intravenous immunoglobulin substitution]. Rev Med Interne. 2006 Dec;27(12):924-6. doi: 10.1016/j.revmed.2006.08.005. Epub 2006 Sep 18. French. PMID 17011081
- [Background] Berger M. Principles of and advances in immunoglobulin replacement therapy for primary immunodeficiency. Immunol Allergy Clin North Am. 2008 May;28(2):413-37, x. doi: 10.1016/j.iac.2008.01.008. PMID 18424340
- [Background] Desai SH, Chouksey A, Poll J, Berger M. A pilot study of equal doses of 10% IGIV given intravenously or subcutaneously. J Allergy Clin Immunol. 2009 Oct;124(4):854-6. doi: 10.1016/j.jaci.2009.07.051. Epub 2009 Sep 19. No abstract available. PMID 19767071
- [Background] Gaspar J, Gerritsen B, Jones A. Immunoglobulin replacement treatment by rapid subcutaneous infusion. Arch Dis Child. 1998 Jul;79(1):48-51. doi: 10.1136/adc.79.1.48. PMID 9771252
- [Background] Haag, S., XIIth Meeting of the European Society for Immunodeficiencies, October 4-7, 2006, Budapest, Hungary. 2012.
- [Background] Shapiro RS. Subcutaneous immunoglobulin: rapid push vs. infusion pump in pediatrics. Pediatr Allergy Immunol. 2013 Feb;24(1):49-53. doi: 10.1111/pai.12026. PMID 23331529
- [Background] Martin A, Lavoie L, Goetghebeur M, Schellenberg R. Economic benefits of subcutaneous rapid push versus intravenous immunoglobulin infusion therapy in adult patients with primary immune deficiency. Transfus Med. 2013 Feb;23(1):55-60. doi: 10.1111/j.1365-3148.2012.01201.x. Epub 2012 Nov 20. PMID 23167310
- [Background] Chapiro, R., XIVth Meeting of the European Society for Immunodeficiencies, October 6-9, 2010, Istanbul, Turkey (R-26). 2010.
- [Background] Nydegger, U.E., Immunoglobulins chap 18 (pp 260-272) in Rossi's principles of transfusion medicine 4th edn Edited by T.L. Simon 2009.
- [Background] Nicolay U, Haag S, Eichmann F, Herget S, Spruck D, Gardulf A. Measuring treatment satisfaction in patients with primary immunodeficiency diseases receiving lifelong immunoglobulin replacement therapy. Qual Life Res. 2005 Sep;14(7):1683-91. doi: 10.1007/s11136-005-1746-x. PMID 16119180
- [Background] Atkinson MJ, Sinha A, Hass SL, Colman SS, Kumar RN, Brod M, Rowland CR. Validation of a general measure of treatment satisfaction, the Treatment Satisfaction Questionnaire for Medication (TSQM), using a national panel study of chronic disease. Health Qual Life Outcomes. 2004 Feb 26;2:12. doi: 10.1186/1477-7525-2-12. PMID 14987333
- [Background] Ware, J., Snow, KK, Kosinski M, Gandek B, SF-36 Health Survey: a manual and interpretation guide. Boston, MA. The Heath Institute, New England Medical Centre. 1993.
- [Background] Cassell EJ. Recognizing suffering. Hastings Cent Rep. 1991 May-Jun;21(3):24-31. No abstract available. PMID 1885294
- [Background] Buchi S, Sensky T. PRISM: Pictorial Representation of Illness and Self Measure. A brief nonverbal measure of illness impact and therapeutic aid in psychosomatic medicine. Psychosomatics. 1999 Jul-Aug;40(4):314-20. doi: 10.1016/S0033-3182(99)71225-9. PMID 10402877
- [Background] Buchi S, Buddeberg C, Klaghofer R, Russi EW, Brandli O, Schlosser C, Stoll T, Villiger PM, Sensky T. Preliminary validation of PRISM (Pictorial Representation of Illness and Self Measure) - a brief method to assess suffering. Psychother Psychosom. 2002 Nov-Dec;71(6):333-41. doi: 10.1159/000065994. PMID 12411768
- [Background] Wouters EJ, Reimus JL, van Nunen AM, Blokhorst MG, Vingerhoets AJ. Suffering quantified? Feasibility and psychometric characteristics of 2 revised versions of the Pictorial Representation of Illness and Self Measure (PRISM). Behav Med. 2008 Summer;34(2):65-78. doi: 10.3200/BMED.34.2.65-78. PMID 18682339
- [Background] Kassardjian CD, Gardner-Nix J, Dupak K, Barbati J, Lam-McCullock J. Validating PRISM (Pictorial Representation of Illness and Self Measure) as a measure of suffering in chronic non-cancer pain patients. J Pain. 2008 Dec;9(12):1135-43. doi: 10.1016/j.jpain.2008.06.016. Epub 2008 Aug 28. PMID 18755635
- [Background] Streffer ML, Buchi S, Morgeli H, Galli U, Ettlin D. PRISM (pictorial representation of illness and self measure): a novel visual instrument to assess pain and suffering in orofacial pain patients. J Orofac Pain. 2009 Spring;23(2):140-6. PMID 19492538
- [Background] Tondury B, Muehleisen B, Ballmer-Weber BK, Hofbauer G, Schmid-Grendelmeier P, French L, Buchi S. The Pictorial Representation of Illness and Self Measure (PRISM) instrument reveals a high burden of suffering in patients with chronic urticaria. J Investig Allergol Clin Immunol. 2011;21(2):93-100. PMID 21462798
- [Background] Wittmann L, Schnyder U, Buchi S. PRISM (Pictorial Representation of Illness and Self Measure): a new method for the assessment of suffering after trauma. J Trauma Stress. 2012 Feb;25(1):94-7. doi: 10.1002/jts.20710. Epub 2012 Jan 25. PMID 22278709
- [Background] Muhleisen B, Buchi S, Schmidhauser S, Jenewein J, French LE, Hofbauer GF. Pictorial Representation of Illness and Self Measure (PRISM): A novel visual instrument to measure quality of life in dermatological inpatients. Arch Dermatol. 2009 Jul;145(7):774-80. doi: 10.1001/archdermatol.2009.121. PMID 19620558
- [Background] Cohen, J. Statistical power analysis for the behavioral sciences (2nd ed.). Hillsdale, NJ : Erlbaum. 1998.
- [Background] Gardulf A, Borte M, Ochs HD, Nicolay U; Vivaglobin Clinical Study Group. Prognostic factors for health-related quality of life in adults and children with primary antibody deficiencies receiving SCIG home therapy. Clin Immunol. 2008 Jan;126(1):81-8. doi: 10.1016/j.clim.2007.06.009. Epub 2007 Oct 26. PMID 17964220
- [Background] Shapiro RS. Why I use subcutaneous immunoglobulin (SCIG). J Clin Immunol. 2013 Jan;33 Suppl 2:S95-8. doi: 10.1007/s10875-012-9853-2. Epub 2012 Dec 21. PMID 23264027
- [Background] Shapiro RS. Subcutaneous immunoglobulin therapy given by subcutaneous rapid push vs infusion pump: a retrospective analysis. Ann Allergy Asthma Immunol. 2013 Jul;111(1):51-5. doi: 10.1016/j.anai.2013.04.015. Epub 2013 May 22. PMID 23806460
- [Background] Orange JS, Grossman WJ, Navickis RJ, Wilkes MM. Impact of trough IgG on pneumonia incidence in primary immunodeficiency: A meta-analysis of clinical studies. Clin Immunol. 2010 Oct;137(1):21-30. doi: 10.1016/j.clim.2010.06.012. Epub 2010 Aug 1. PMID 20675197
- [Background] Quinti I, Soresina A, Guerra A, Rondelli R, Spadaro G, Agostini C, Milito C, Trombetta AC, Visentini M, Martini H, Plebani A, Fiorilli M; IPINet Investigators. Effectiveness of immunoglobulin replacement therapy on clinical outcome in patients with primary antibody deficiencies: results from a multicenter prospective cohort study. J Clin Immunol. 2011 Jun;31(3):315-22. doi: 10.1007/s10875-011-9511-0. Epub 2011 Mar 2. PMID 21365217